CLINICAL TRIAL: NCT05627089
Title: Rheumatoid Arthritis and Myositis Cohort
Status: Withdrawn | Type: Observational
Why Stopped: Decided not to move forward
Sponsor: Attune Health Research, Inc. (Industry)
Collaborators: ONCOtracker Inc (Industry)
Responsible Party: Principal Investigator, Swamy Venuturupalli, Principal Investigator, Attune Health Foundation
Other Study IDs: RAMC2022
Record Dates: First submitted 2022-11-09; First posted 2022-11-25 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Rheumatoid Arthritis; Myositis
Keywords: Intestinal Microbiome; Immune cells; Cytokines; Rheumatoid Arthritis; Myositis; Autoimmune disease; Immunosuppressive medication; Diet; Disease Activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Myositis; Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, serum, plasma, urine, stool, synovial tissue, skin tissue, muscle tissue, extract DNA and RNA, endoscopy aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Rheumatoid Arthritis and/or Myositis: All patients 18 years or older who have been diagnosed with Rheumatoid Arthritis according to the 2010 ACR/EULAR Classification Criteria.
  All patients 18 years or older who have been diagnosed with Myositis according to the 2017 European League Against Rheumatism/American College of Rheumatology Classification Criteria for Adult and Juvenile Idiopathic Inflammatory Myopathies Classification Criteria.

SUMMARY:
The primary objective of this research is to establish a well characterized clinical and longitudinal cohort for individuals with Rheumatoid Arthritis (RA) and Myositis to create a place to maintain blood, urine, stool specimens, excess tissue from procedures, and clinical data, which may be accessed for future research purposes.

Specific research objectives of this cohort include:

1. Observe the response that immunosuppressive medications have on the immune cell population and cytokines in individuals with RA or Myositis.
2. Observe the role that the intestinal microbiome has on the immune cell population and cytokines in individuals with RA or Myositis.
3. Observe the connection between intestinal inflammation has on the immune cell population and cytokines in individuals with RA or Myositis.

DETAILED DESCRIPTION:
Autoimmune diseases are together the third most common type of disease that affect individuals in the United States. In 2005 the National Institute of Health estimated that 23.5 million people have an autoimmune condition. Previously considered to be rare, epidemiological studies have shown that there are nearly 100 different autoimmune diseases. Examples include organ specific autoimmune disease such as Primary Biliary Cirrhosis (PBC), or Systematic Lupus Erythematosus, which reflects immunological dysfunction involving multiple organs. As the prevalence and incidence of autoimmune diseases continue to rise, it creates a burden on individuals, their families, and society. The burden is noticeable through medical costs, diminished quality of life, and loss of productivity. The burden of this disease demands a comprehensive treatment that includes overall wellness.

The human gastrointestinal tract is home to trillions of microorganisms including bacteria, viruses, fungi, and protozoa, which together are referred to as the gut microbiome. Research in recent years has underlined that the microorganisms can influence varying physiological aspects such as the immune system, metabolism, and behavior. The microbiome has further been implicated in the pathogenesis of autoimmune diseases. In Systematic Lupus Erythematosus for example, modifications in the intestinal flora have been documented while changes in gut commensal and periodontal diseases have been brought forth as factors for consideration in the development of Rheumatoid Arthritis. Similarly, autoimmune diseases such as Systematic Sclerosis, Sjogren's Syndrome, and Anti-phospholipid Syndrome have been noted to share alterations in the gut microbiome.

Emerging research on the gut microbiome has demonstrated that diet plays a critical role in the make-up of gut microbiome and several experiments have shown that dietary modifications can prompt significant changes in the gut microbial composition. However, little is presently understood about the precise mechanisms and unique interactions between the gut microbiome, diet, and the pathogenesis of autoimmune diseases.

To investigate the triangular link between a patient's diet, their microbiome, and their disease activity, the investigators are seeking to establish a registry to track patients with autoimmune disease diagnoses. Furthermore, the investigators are looking to track the changes in the microbiome, diet, and disease progression as patients are introduced and sustained on medication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years or older
* Diagnosed RA by a rheumatologist determined by the 2010 ACR/EULAR Classification Criteria.
* Diagnosed Myositis by a rheumatologist determined by the 2017 American College of Rheumatology Classification Criteria for Adult and Juvenile Idiopathic Inflammatory Myopathies
* Able to read and write in English or Spanish

Exclusion Criteria:

* Subject is less than 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients seen with Rheumatoid Arthritis or Myositis who are at least 18 years of age will be eligible for the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2033-01-01 (Estimated); Study Completion 2035-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in IL-1, IL-6, CXCL10 and Immune Cell Population due to Immunosuppressive Medication | 1 year
  Observe the response that immunosuppressive medications have on the immune cell population and cytokines in individuals with RA or Myositis.
Change in IL-1, IL-6, CXCL10 and Immune Cell Population in response to Intestinal Microbiome | 1 year
  Observe the role that the intestinal microbiome has on the immune cell population and cytokines in individuals with RA or Myositis.
Change in IL-1, IL-6, CXCL10 and Immune Cell Population in response to Intestinal Inflammation | 1 year
  Observe the connection between intestinal inflammation has on the immune cell population and cytokines in individuals with RA or Myositis.

SECONDARY OUTCOMES:
Change in IL-1, IL-6, CXCL10 and Immune Cell Population due to Immunosuppressive Medication | 10 years
  Observe the response that immunosuppressive medications have on the immune cell population and cytokines in individuals with RA or Myositis.
Change in IL-1, IL-6, CXCL10 and Immune Cell Population due to changes in the intestinal microbiome | 10 years
  Observe the response that immunosuppressive medications have on the immune cell population and cytokines in individuals with RA or Myositis.
Change in IL-1, IL-6, CXCL10 and Immune Cell Population due to Intestinal Inflammation | 10 years
  Observe the connection between intestinal inflammation has on the immune cell population and cytokines in individuals with RA or Myositis.

REFERENCES:
- [Background] Bethesda. National Institutes of Health Autoimmune Disease Coordinating Committee Report. The Institutes, 2002.
- [Background] Services USDoHaH. Progress in Autoimmune Diseases and Research. National Institutes of Health: The autoimmune Diseases Coordinating Committee, 2005:1-126.
- [Background] Wang L, Wang FS, Gershwin ME. Human autoimmune diseases: a comprehensive update. J Intern Med. 2015 Oct;278(4):369-95. doi: 10.1111/joim.12395. Epub 2015 Jul 25. PMID 26212387
- [Background] Xu J, Yang Y. Gut microbiome and its meta-omics perspectives: profound implications for cardiovascular diseases. Gut Microbes. 2021 Jan-Dec;13(1):1936379. doi: 10.1080/19490976.2021.1936379. PMID 34170211
- [Background] De Luca F, Shoenfeld Y. The microbiome in autoimmune diseases. Clin Exp Immunol. 2019 Jan;195(1):74-85. doi: 10.1111/cei.13158. PMID 29920643
- [Background] Singh RK, Chang HW, Yan D, Lee KM, Ucmak D, Wong K, Abrouk M, Farahnik B, Nakamura M, Zhu TH, Bhutani T, Liao W. Influence of diet on the gut microbiome and implications for human health. J Transl Med. 2017 Apr 8;15(1):73. doi: 10.1186/s12967-017-1175-y. PMID 28388917
- [Background] Vieira SM, Pagovich OE, Kriegel MA. Diet, microbiota and autoimmune diseases. Lupus. 2014 May;23(6):518-26. doi: 10.1177/0961203313501401. PMID 24763536
- [Background] Anderson J, Caplan L, Yazdany J, Robbins ML, Neogi T, Michaud K, Saag KG, O'Dell JR, Kazi S. Rheumatoid arthritis disease activity measures: American College of Rheumatology recommendations for use in clinical practice. Arthritis Care Res (Hoboken). 2012 May;64(5):640-7. doi: 10.1002/acr.21649. PMID 22473918
- [Result] Fransen J, van Riel PL. The Disease Activity Score and the EULAR response criteria. Rheum Dis Clin North Am. 2009 Nov;35(4):745-57, vii-viii. doi: 10.1016/j.rdc.2009.10.001. PMID 19962619
- [Result] Rider LG, Aggarwal R, Machado PM, Hogrel JY, Reed AM, Christopher-Stine L, Ruperto N. Update on outcome assessment in myositis. Nat Rev Rheumatol. 2018 May;14(5):303-318. doi: 10.1038/nrrheum.2018.33. Epub 2018 Apr 12. PMID 29651119
- [Result] Instruments available for use in Assessment Center . Secondary Instruments available for use in Assessment Center. https://www.assessmentcenter.net/documents/InstrumentLibrary.pdf.
- [Result] Deyo RA, Katrina Ramsey, Buckley DI, Michaels L, Kobus A, Eckstrom E, Forro V, Morris C. Performance of a Patient Reported Outcomes Measurement Information System (PROMIS) Short Form in Older Adults with Chronic Musculoskeletal Pain. Pain Med. 2016 Feb;17(2):314-24. doi: 10.1093/pm/pnv046. PMID 26814279
- [Result] Bigaard J, Frederiksen K, Tjonneland A, Thomsen BL, Overvad K, Heitmann BL, Sorensen TI. Waist circumference and body composition in relation to all-cause mortality in middle-aged men and women. Int J Obes (Lond). 2005 Jul;29(7):778-84. doi: 10.1038/sj.ijo.0802976. PMID 15917857
- [Result] Konijn NP, van Tuyl LH, Bultink IE, Lems WF, Earthman CP, van Bokhorst-de van der Schueren MA. Making the invisible visible: bioelectrical impedance analysis demonstrates unfavourable body composition in rheumatoid arthritis patients in clinical practice. Scand J Rheumatol. 2014;43(4):273-8. doi: 10.3109/03009742.2013.852239. Epub 2014 Feb 7. PMID 24797672
- [Result] Chen YM, Chen HH, Hsieh CW, Hsieh TY, Lan JL, Chen DY. A close association of body cell mass loss with disease activity and disability in Chinese patients with rheumatoid arthritis. Clinics (Sao Paulo). 2011;66(7):1217-22. doi: 10.1590/s1807-59322011000700016. PMID 21876977
- [Result] Sciences NCIDoCCP. DHQIII Diet History Questionnaire Secondary DHQIII Diet History Questionnaire https://epi.grants.cancer.gov/dhq3/.
- [Result] Thompson FE, Subar AF, Brown CC, Smith AF, Sharbaugh CO, Jobe JB, Mittl B, Gibson JT, Ziegler RG. Cognitive research enhances accuracy of food frequency questionnaire reports: results of an experimental validation study. J Am Diet Assoc. 2002 Feb;102(2):212-25. doi: 10.1016/s0002-8223(02)90050-7. PMID 11846115
- [Result] Subar AF, Thompson FE, Kipnis V, Midthune D, Hurwitz P, McNutt S, McIntosh A, Rosenfeld S. Comparative validation of the Block, Willett, and National Cancer Institute food frequency questionnaires : the Eating at America's Table Study. Am J Epidemiol. 2001 Dec 15;154(12):1089-99. doi: 10.1093/aje/154.12.1089. PMID 11744511
- [Result] Subar AF, Kipnis V, Troiano RP, Midthune D, Schoeller DA, Bingham S, Sharbaugh CO, Trabulsi J, Runswick S, Ballard-Barbash R, Sunshine J, Schatzkin A. Using intake biomarkers to evaluate the extent of dietary misreporting in a large sample of adults: the OPEN study. Am J Epidemiol. 2003 Jul 1;158(1):1-13. doi: 10.1093/aje/kwg092. PMID 12835280